CLINICAL TRIAL: NCT01597453
Title: NOR-SYS: The Norwegian Stroke in the Young Study Young Ischemic Stroke and Family Risk Factors
Brief Title: NOR-SYS: The Norwegian Stroke in the Young Study
Acronym: NOR-SYS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/74
Record Dates: First submitted 2012-05-02; First posted 2012-05-14 (Estimated); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Death; Carotid Artery Disease; Cardiovascular Disease; Peripheral Artery Disease
Keywords: Young ischemic stroke; Families; Long-term follow-up
MeSH Terms: conditions — Death; Carotid Artery Diseases; Cardiovascular Diseases; Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: Inclusion was completed in 2015, and the 5-year follow-up phase was completed in july 2021. The planned 10-year follow-up has not been possible due to the covid pandemia. A final 15 year follow-up was originally planned, and would start in 2025.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lifestyle counseling (Other): There are no different arms, NOR-SYS is an observational study
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: Lifestyle counseling — Ultrasound examinations of carotid arteries, aorta abdominalis, femoral arteries and lifestyle counseling
  Other Names: NOR-SYS

SUMMARY:
NOR-SYS is a clinical research program about young ischemic stroke patients from 15 to 60 years. Patients, partners and the couple´s adult children who are at least 18 years old, are all invited to ultrasound examinations due to a standardized protocol.

Parents of patients and partners are invited to return their answers of standardized questionnaires about clinical ischemic events such as stroke, angina or myocardial infarction or peripheral artery disease.

Study inclusion time of patients and their families is 5 years. A biobank is build from samples from patients, partners and adult children. Clinical follow-ups for patients and partners are planned after 5, 10 and 15 years. Clinical follow-ups for adult children are planned after 10 and 20 years.

Hypotheses:

What do patients know about their parents clinical ischemic events? How much established pathology in arteries do we find by a standardized ultrasound protocol at the time of ischemic stroke at a young age? Differences concerning risk factors and ultrasound findings between patients and partners? Differences between children from families with several ischemic events among parents and grandparents vs. children from families without ischemic events? Biochemical markers related to ultrasound findings and artery disease.

DETAILED DESCRIPTION:
Equal examinations for patients, partners and adult children are:

* Standardized questionnaires
* Extracranial duplexsonography
* Duplexsonography of the abdominal aorta
* Duplexsonography of femoral arteries
* Duplexsonography of epicardial, intrabdominal and subcutaneous fat
* Peripheral ultrasound, Ankle-arm index
* ECG
* Blood pressure measurement
* BMI and Waist-hip ratio
* Blood samples

ELIGIBILITY:
Inclusion Criteria:

* Documented ischemic stroke at age from 15 up to 60 years

Exclusion Criteria:

* Stroke as end-of-life event among patients with cancer or other life-threatening disease
* Stroke caused by trauma

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1062 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 15 years for patients and partners and 20 years for offspring
  Outcome measure is assessed every five years.

SECONDARY OUTCOMES:
Arterial events (recurrent stroke or transitory ischemic attack, myocardial infarction or angina, peripheral artery disease | 15 years for patients and partners and 20 years for offspring
  Outcome measure is assessed every five years.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Waje-Andreassen, MD, PhD, Principal Investigator — Haukeland UH
Locations (1):
- Dep. of Neurology, Bergen, Norway

REFERENCES:
- [Derived] Jibril KA, Kuiper KJ, Nawaz B, Naess H, Fromm A, Oygarden H, Sand KM, Meijer R, Mohamed Ali A, Larsen TH, Bleie O, Skaar E, Waje-Andreassen U, Saeed S. Burden of Coronary Artery Disease as a Predictor of New Vascular Events and Mortality in Patients With Ischemic Stroke: Insights From the Norwegian Stroke in the Young Study. J Am Heart Assoc. 2025 Mar 18;14(6):e038899. doi: 10.1161/JAHA.124.038899. Epub 2025 Mar 13. PMID 40079310
- [Derived] Oftedal A, Gerdts E, Waje-Andreassen U, Fromm A, Naess H, Linde A, Saeed S. Prevalence and covariates of uncontrolled hypertension in ischemic stroke survivors: the Norwegian stroke in the young study. Blood Press. 2018 Jun;27(3):173-180. doi: 10.1080/08037051.2018.1425827. Epub 2018 Jan 15. PMID 29334265
- [Derived] Oygarden H, Fromm A, Sand KM, Kvistad CE, Eide GE, Thomassen L, Naess H, Waje-Andreassen U. A Family History of Stroke Is Associated with Increased Intima-Media Thickness in Young Ischemic Stroke - The Norwegian Stroke in the Young Study (NOR-SYS). PLoS One. 2016 Aug 9;11(8):e0159811. doi: 10.1371/journal.pone.0159811. eCollection 2016. PMID 27504830
- [Derived] Oygarden H, Fromm A, Sand KM, Eide GE, Thomassen L, Naess H, Waje-Andreassen U. Stroke patients' knowledge about cardiovascular family history - the Norwegian Stroke in the Young Study (NOR-SYS). BMC Neurol. 2015 Mar 12;15:30. doi: 10.1186/s12883-015-0276-6. PMID 25884546
- [Derived] Saeed S, Waje-Andreassen U, Fromm A, Oygarden H, Kokorina MV, Naess H, Gerdts E. Early vascular aging in young and middle-aged ischemic stroke patients: the Norwegian Stroke in the Young Study. PLoS One. 2014 Nov 18;9(11):e112814. doi: 10.1371/journal.pone.0112814. eCollection 2014. PMID 25405619
- [Derived] Fromm A, Haaland OA, Naess H, Thomassen L, Waje-Andreassen U. Risk factors and their impact on carotid intima-media thickness in young and middle-aged ischemic stroke patients and controls: the Norwegian Stroke in the Young Study. BMC Res Notes. 2014 Mar 26;7:176. doi: 10.1186/1756-0500-7-176. PMID 24669965
- [Derived] Fromm A, Thomassen L, Naess H, Meijer R, Eide GE, Krakenes J, Vedeler CA, Gerdts E, Larsen TH, Kuiper KK, Laxdal E, Russell D, Tatlisumak T, Waje-Andreassen U. The Norwegian Stroke in the Young Study (NOR-SYS): rationale and design. BMC Neurol. 2013 Jul 17;13:89. doi: 10.1186/1471-2377-13-89. PMID 23865483